CLINICAL TRIAL: NCT04377568
Title: A Randomized, Multicentered, Open-label Phase 2 Clinical Trial of the Safety and Efficacy of Human Coronavirus- Immune Convalescent Plasma for the Treatment of COVID-19 Disease in Hospitalized Children
Brief Title: Efficacy of Human Coronavirus-immune Convalescent Plasma for the Treatment of COVID-19 Disease in Hospitalized Children
Acronym: CONCOR-KIDS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no enrollment
Sponsor: The Hospital for Sick Children (Other)
Collaborators: C17 Council (regulatory sponsor) (Unknown)
Responsible Party: Principal Investigator, Julia Upton, Staff Physician, Allergy and Immunology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000070143
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hospitalized Children; Covid-19 Infection
Keywords: covid-19; hospitalized children; convalescent plasma therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either standard of care (SoC) products (control) or COVID-19 convalescent plasma (C19-CP) plus standard of care while being hospitalized for COVID-19 (ratio 1:2). The intervention will consist of a single transfusion of convalescent plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma + Standard of Care (C19-CP + SoC) (Experimental): Participants will receive COVID-19 convalescent plasma (C19-CP) plus standard of care while being hospitalized for COVID-19.
  Interventions: Biological: Convalescent plasma (CP)
- Standard of Care (SoC) (No Intervention): Participants will receive standard of care while being hospitalized for COVID-19.

INTERVENTIONS:
Biological: Convalescent plasma (CP) — Participants will receive one infusion of convalescent plasma proportional to their weight (10 mL/kg), up to a maximum of 500 mL
  Arms: Convalescent Plasma + Standard of Care (C19-CP + SoC)

SUMMARY:
This is a multicentered, open-label, randomized controlled Phase 2 trial to evaluate the safety and efficacy of providing human coronavirus-immune convalescent plasma as treatment for COVID-19 disease in hospitalized children in the context of the COVID-19 pandemic.

DETAILED DESCRIPTION:
SARS-CoV-2 viral infection resulting in COVID-19 disease has recently been designated by the World Health Organization as a global pandemic. Outbreak forecasting and mathematical models suggest that the number of COVID-19 cases will continue to rise over the coming weeks and months. There is an urgent public health need for rapid development of novel interventions. This protocol aims to use passive antibody therapy via convalescent plasma from SARS-CoV-2-infected patients who have developed antibody immunity, COVID-19 convalescent plasma (C19-CP), as treatment for hospitalized children with COVID-19 disease at pediatric academic hospitals across Canada. The unknown role for convalescent plasma in treating COVID-19 necessitates further study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 to <19 years old
2. Hospitalized with symptoms compatible with COVID-19 illness
3. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen prior to randomization.
4. ABO compatible convalescent plasma available

Exclusion Criteria:

1. Onset of symptoms began >12 days before screening
2. History of adverse reactions to blood products or other contraindication to transfusion
3. Refusal of plasma for religious or other reasons
4. Acute heart failure with fluid overload
5. Any condition or diagnosis, that could in the opinion of the Site Principal Investigator interfere with the participant's ability to comply with study instructions, or put the participant at risk
6. Anticipated discharge within 24 hours

Note: The intent of this exclusion criteria is to only include participants with acute COVID-19 infections. This protocol is not intended to include participants with post-infectious complications. In cases where the distinction is not clear, participant eligibility will be discussed with the study steering committee prior to enrollment.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery | at day 30
  defined in the last 24 hours as normal respiratory and heart rate (or return to baseline, absence of fever, absence of low blood pressure, oxygen saturation greater than 94% or room air (or return to baseline), no need for intravenous fluids (or return to baseline)

SECONDARY OUTCOMES:
Combined mortality/intubation | at 30 day
  Proportion of patients experiencing death in hospital (Yes/No) 30 days
Respiratory status-1 | at 30 days
  Proportion of patients experiencing Intubation (Yes/No)
Respiratory status-2 | time from admission to intubation
  time to intubation
Respiratory status-3 | from admission to day 30 of hospitalization
  Mean number of ventilator-free days in 30 days
respiratory status -4 | from admission to day 30 of hospitalization
  Mean number of ventilator days in 30 days
respiratory status -5 | from admission to day 30 of hospitalization
  The number of oxygen free days in the first 30 days or the incidence and duration of new oxygen use during the trial, defined as oxygen use that was not present at time of randomization but occurs subsequently
respiratory status-6 | at 30 days
  The proportion of patients needing ECMO in 30 days
Mortality 1a | at 30 days
  Time to in-hospital death censored
Mortality 1b | at 90 days
  Time to in-hospital death censored
Mortality 2a | at 30 days
  Proportion of patients with Survival status
Mortality 2b | at 90 days
  Proportion of patients with Survival status
Care and Critical Care | at 30 days
  Length of hospitalization and stay in the ICU
organ systems: renal | up to 365 days
  The proportion of patients needing renal replacement therapy
organ systems: cardiac | up to 365 days
  The proportion of patients developing myocarditis
Transfusion-associated adverse events (AE) | up to 365 days
  The proportion of patients developing adverse events to the treatment arm, C19-CP as assessed by Proposed Standard definitions for surveillance of non-infectious adverse transfusion reactions.
Safety of the intervention | up to 365 days
  cumulative incidence of severe and life-threatening AEs and severe AEs
organ systems: multi-system inflammatory disease | up to 365 days
  The proportion of patients developing multi-system inflammatory disease

OTHER OUTCOMES:
Virological measures 1 | at day 3
  Proportion of patients with negative virology
Virological measures 3 | at day 10
  Proportion of patients with negative virology
Virological measures 4 | at day 15
  Proportion of patients with negative virology
Modulation of biomarkers | up to 365 days
  Exploratory analysis of biomarker differences between groups
Resolution of fever | hours
  Time to fever resolution (no longer requiring fever management)
Presence and titres levels | at day 30
  Presence and titres of IgG, IgA antibodies and neutralizing antibody titres in C19-CP group on the primary outcome and other outcomes.
Functional measure 1 | up to 365 days
  efficacy of C19-CP on respiratory measures using pediatric validated dyspnea (breathlessness) scales
Functional measure 2 | up to 365 days
  Evaluate the efficacy of C19-CP on quality of life (QOL) measures using Validated QOL scores (Eq-5D)
Functional measure 3 | up to 365 days
  Evaluate the efficacy of C19-CP on rehospitalization after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Julia Upton, MD, MPH, Study Chair — The Hospital for Sick Children; Kathy Brodeur-Robb, Study Director — C17 Council (regulatory sponsor)
Locations (13):
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Winnipeg Children's Hospital, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - McGill Univ Health Ctr - Montreal Children's Hospital, Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan